CLINICAL TRIAL: NCT05522010
Title: Dynamic Cervical Implant (DCI) Versus Anterior Cervical Discectomy And Fusion(ACDF) For The Treatment Of Single-Level Cervical Degenerative Disc Disease (DDD): An RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelrahman Saleh El Attar, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cervical Degenerative Disease
Record Dates: First submitted 2022-08-19; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Cervical Degenerative Disc Disease
Keywords: Cervical Degenerative Disc Disease; Dynamic Cervical Implant; Anterior Cervical Discectomy And Fusion

STUDY DESIGN:
Intervention Model Description: A calculated minimum sample of 50 patients with single or multiple symptomatic cervical DDD with radiculopathy and\or myelopathy not responding to non-surgical management will be needed. The sample will be randomly assigned for one of two equal groups (Group I (n=25); will undergo ACDF and Group II (n=25) will undergo DCI to detect an effect size of 0.42 in the rate of adjacent segment degeneration (main clinical and radiological outcomes), with an error probability of 0.05 and 80%
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (1) (ACDF) (Active Comparator): All patients on this group will undergo Anterior Cervical Discectomy And Fusion
  Interventions: Procedure: Cervical spine surgery
- Group (2) (DCI) (Active Comparator): All patients on this group will undergo Dynamic Cervical Implant
  Interventions: Procedure: Cervical spine surgery

INTERVENTIONS:
Procedure: Cervical spine surgery — A standard anterior approach was made with discectomy sparing the cartilage, and with foraminal decompression. Complete excision of the posterior longitudinal ligament was routinely performed to complete neural decompression. Trial inserters were used to identify the proper implant size. Device under sizing may lead to poor ﬁxation and implant migration. The largest possible device that can be safely placed should be selected to maximize device- endplate contact and to gain support from the apophyseal rim. The teeth of the implant were optimally ﬁxated to the endplate via Caspar pin compression following device insertion. The device may be replaced or changed using the same insertion instrument if ﬁnal imaging demonstrated suboptimal positioning. Rinsing the implanted disc space removes rests of blood and bone dust, all potentially promoting HO

SUMMARY:
TO Compare The Clinical And Radiographic Outcomes of DCI VS ACDF For The Treatment Of Single-Level Cervical Degenerative Disc Disease (DDD)

DETAILED DESCRIPTION:
Anterior cervical discectomy and fusion (ACDF) is an effective and safe treatment for patients with radiculopathy and myelopathy. However, in the untreated levels adjacent to a fusion, increased motion and elevated intradiscal pressures have been reported. Some investigators have postulated that these changes may lead to an increased risk of adjacent segment degeneration (ASD). Limitations and problems with ACDF have led some investigators to explore the motion-preserving surgeries, such as cervical total disk replacement (TDR). Although TDR has been shown to reduce adjacent-level intra discal pressures and provide a more physiological overall cervical but also index- and adjacent-level range of motion (ROM) while maintaining sagittal alignment. Recent studies have also highlighted the potential limitations of TDR. Dynamic cervical implant (DCI) is a type of anterior decompression and cervical non-fusion implant that was initially conceived as a method to combine the potential advantages of fusion and TDR. The DCI is intended to provide controlled, limited flexion and extension-the primary motions in the sub axial cervical spine-that is greater than that seen with fusion, but less than that achieved with TDR .

ELIGIBILITY:
Inclusion Criteria:

* Single or multiple symptomatic cervical DDD with radiculopathy and\or mylopathy not responding to non-surgical management
* Age older than 18 years

Exclusion Criteria:

1. ossification of posterior longitudinal ligament
2. facet arthritis
3. lack of motion or instability at the level of surgery
4. fracture
5. infection
6. tumors
7. osteoprosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-25 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Radiological outcome | At 1 year follow up.
  MRI grading for the degree of ASD (Mario Matsumato grading)

SECONDARY OUTCOMES:
Clinical outcome | At 3 month .
  1-Neck Disability Index (NDI) : 10 item score from 0 to 5 maximum score is 50 , high score is worse
Radiological outcome (Plain x-ray) | at 6 month.
  1- Cervical sagittal alignment C2 to C7 (Cobb angle)
  5-implant fusion described as a less than 1-mm motion between the tips of the spinous processes in dynamic radiographs and/or the presence of bridging bony trabeculae.
Radiological outcome (MSCT) | At 1 year .
  1-implant fusion
clinical outcome | At 3 month .
  Visual analogue scale (VAS) scores for neck and arm from 0 to 10 score , the higher score is worse
radiological outcome | at 6 month .
  2- Range of motion (ROM) using Cobb method for cervical spine and functional spine unit of treated segment

REFERENCES:
- [Background] Irwin ZN, Hilibrand A, Gustavel M, McLain R, Shaffer W, Myers M, Glaser J, Hart RA. Variation in surgical decision making for degenerative spinal disorders. Part II: cervical spine. Spine (Phila Pa 1976). 2005 Oct 1;30(19):2214-9. doi: 10.1097/01.brs.0000181056.76595.f7. PMID 16205349
- [Background] Fuller DA, Kirkpatrick JS, Emery SE, Wilber RG, Davy DT. A kinematic study of the cervical spine before and after segmental arthrodesis. Spine (Phila Pa 1976). 1998 Aug 1;23(15):1649-56. doi: 10.1097/00007632-199808010-00006. PMID 9704371
- [Background] Hilibrand AS, Yoo JU, Carlson GD, Bohlman HH. The success of anterior cervical arthrodesis adjacent to a previous fusion. Spine (Phila Pa 1976). 1997 Jul 15;22(14):1574-9. doi: 10.1097/00007632-199707150-00009. PMID 9253091
- [Background] Shao MM, Chen CH, Lin ZK, Wang XY, Huang QS, Chi YL, Wu AM. Comparison of the more than 5-year clinical outcomes of cervical disc arthroplasty versus anterior cervical discectomy and fusion: A protocol for a systematic review and meta-analysis of prospective randomized controlled trials. Medicine (Baltimore). 2016 Dec;95(51):e5733. doi: 10.1097/MD.0000000000005733. PMID 28002345
- [Background] Coric D, Kim PK, Clemente JD, Boltes MO, Nussbaum M, James S. Prospective randomized study of cervical arthroplasty and anterior cervical discectomy and fusion with long-term follow-up: results in 74 patients from a single site. J Neurosurg Spine. 2013 Jan;18(1):36-42. doi: 10.3171/2012.9.SPINE12555. Epub 2012 Nov 9. PMID 23140129
- [Background] Zou S, Gao J, Xu B, Lu X, Han Y, Meng H. Anterior cervical discectomy and fusion (ACDF) versus cervical disc arthroplasty (CDA) for two contiguous levels cervical disc degenerative disease: a meta-analysis of randomized controlled trials. Eur Spine J. 2017 Apr;26(4):985-997. doi: 10.1007/s00586-016-4655-5. Epub 2016 Jun 17. PMID 27314663
- [Background] Gornet MF, Lanman TH, Burkus JK, Hodges SD, McConnell JR, Dryer RF, Copay AG, Nian H, Harrell FE Jr. Cervical disc arthroplasty with the Prestige LP disc versus anterior cervical discectomy and fusion, at 2 levels: results of a prospective, multicenter randomized controlled clinical trial at 24 months. J Neurosurg Spine. 2017 Jun;26(6):653-667. doi: 10.3171/2016.10.SPINE16264. Epub 2017 Mar 17. PMID 28304237
- [Background] Radcliff K, Coric D, Albert T. Five-year clinical results of cervical total disc replacement compared with anterior discectomy and fusion for treatment of 2-level symptomatic degenerative disc disease: a prospective, randomized, controlled, multicenter investigational device exemption clinical trial. J Neurosurg Spine. 2016 Aug;25(2):213-24. doi: 10.3171/2015.12.SPINE15824. Epub 2016 Mar 25. PMID 27015130
- [Background] Wu TK, Wang BY, Meng Y, Ding C, Yang Y, Lou JG, Liu H. Multilevel cervical disc replacement versus multilevel anterior discectomy and fusion: A meta-analysis. Medicine (Baltimore). 2017 Apr;96(16):e6503. doi: 10.1097/MD.0000000000006503. PMID 28422837
- [Background] Lu VM, Zhang L, Scherman DB, Rao PJ, Mobbs RJ, Phan K. Treating multi-level cervical disc disease with hybrid surgery compared to anterior cervical discectomy and fusion: a systematic review and meta-analysis. Eur Spine J. 2017 Feb;26(2):546-557. doi: 10.1007/s00586-016-4791-y. Epub 2016 Sep 27. PMID 27679431
- [Background] Kelly MP, Eliasberg CD, Riley MS, Ajiboye RM, SooHoo NF. Reoperation and complications after anterior cervical discectomy and fusion and cervical disc arthroplasty: a study of 52,395 cases. Eur Spine J. 2018 Jun;27(6):1432-1439. doi: 10.1007/s00586-018-5570-8. Epub 2018 Mar 31. PMID 29605899
- [Background] Pickett GE, Sekhon LH, Sears WR, Duggal N. Complications with cervical arthroplasty. J Neurosurg Spine. 2006 Feb;4(2):98-105. doi: 10.3171/spi.2006.4.2.98. PMID 16506475
- [Background] Li Z, Yu S, Zhao Y, Hou S, Fu Q, Li F, Hou T, Zhong H. Clinical and radiologic comparison of dynamic cervical implant arthroplasty versus anterior cervical discectomy and fusion for the treatment of cervical degenerative disc disease. J Clin Neurosci. 2014 Jun;21(6):942-8. doi: 10.1016/j.jocn.2013.09.007. Epub 2013 Nov 4. PMID 24411326
- [Background] Wang L, Song YM, Liu LM, Liu H, Li T. Clinical and radiographic outcomes of dynamic cervical implant replacement for treatment of single-level degenerative cervical disc disease: a 24-month follow-up. Eur Spine J. 2014 Aug;23(8):1680-7. doi: 10.1007/s00586-014-3180-7. Epub 2014 Jan 29. PMID 24474644